CLINICAL TRIAL: NCT00429871
Title: A Multicenter Randomized Comparative Study of Docetaxel Plus Epirubicin Versus Docetaxel Plus Capecitabine Combinations as First Line Treatment of Metastatic Breast Cancer
Brief Title: Randomized Phase III Trial With Docetaxel Plus Epirubicine Versus Docetaxel Plus Capecitabine for Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: D.Mavrudis, Hellenic Oncology Research Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT/02.09
Record Dates: First submitted 2007-01-31; First posted 2007-02-01 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Breast Cancer
Keywords: Metastatic breast cancer;; First line chemotherapy;; Docetaxel;; Epirubicin;; Capecitabine
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Capecitabine; Epirubicin

ARMS (2):
- 1 (Experimental): DF
  Interventions: Drug: Docetaxel; Drug: Epirubicin
- 2 (Experimental): DC
  Interventions: Drug: Capecitabine; Drug: Docetaxel

INTERVENTIONS:
Drug: Docetaxel — Docetaxel at the dose of 75mg/m2 IV on day 1 every 3 weeks for 6 consecutive cycles
  Other Names: Taxotere
  Arms: 1
Drug: Capecitabine — Capecitabine 950 mg/m2 orally twice a day on days 1-14 every 3 weeks for 6 consecutive cycles
  Other Names: Xeloda
  Arms: 2
Drug: Epirubicin — Epirubicin at the dose of 75mg/m2 IV on day 1 every 3 weeks for 6 consecutive cycles
  Other Names: Farmorubicin
  Arms: 1
Drug: Docetaxel — Docetaxel at the dose of 75mg/m2 IV on day 1 every 3 weeks for 6 consecutive cycles
  Other Names: Taxotere
  Arms: 2

SUMMARY:
The combination of docetaxel+epirubicin is highly effective and well tolerated as first line treatment in patients with metastatic breast cancer (MBC). Capecitabine is an active drug in women with MBC pretreated with taxane and anthracycline. Docetaxel increases the intracellular levels of thymidilate phosphorylase and thus is synergistic with capecitabine. The combination of docetaxel plus capecitabine is highly active and superior to docetaxel monotherapy in women with MBC pretreated with an anthracycline

DETAILED DESCRIPTION:
This trial will compare the efficacy of docetaxel plus epirubicin versus docetaxel plus capecitabine combinations as first line treatment in women with MBC

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically- confirmed metastatic breast adenocarcinoma.
* No previous chemotherapy treatment for metastatic disease.
* No previous anthracycline treatment except as adjuvant therapy at least one year before.
* Age 19-75 years old
* Presence of measurable disease
* Performance status 0-2 (WHO)
* Adequate cardiac function (LVEF >50%) without a recent (within 6 months) history of myocardial infraction and/or unstable or uncontrolled angina.
* Adequate bone marrow(absolute neutrophil count >1500/mm3, platelet count >100.000/mm3, hemoglobin >10gr/mm3), liver (bilirubin <1.5 times upper limit of normal and SGOT/SGPT <2 times upper limit of normal) and renal function (creatinine <2mg/dl).
* No previous radiotherapy to more than 25% of marrow-containing bones.
* Written informed consent

Exclusion Criteria:

* Active brain metastases.
* Psychiatric illness or social situation that would preclude study compliance
* Other concurrent uncontrolled illness.
* Other invasive malignancy within the past 5 years except of nonmelanoma skin cancer.
* Positive pregnancy for premenopausal women.
* Concurrent antineoplastic treatment e.g. hormonal therapy

Ages: 19 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2002-05; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Compare the time to tumor progression between the two treatment arms | 1 year

SECONDARY OUTCOMES:
Overall survival | 1 year
Toxicity profile between the two treatment arms | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Mavrudis, MD, Principal Investigator — University Hospital of Crete, Dep of Medical Oncology
Locations (10):
- Greece (10):
  - University Hospital of Heraklion, Heraklion, Crete
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - "IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - "Marika Iliadis" Hospital of Athens, Dep of Medical Oncology, Athens
  - 401 Military Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens, Athens
  - State General Hospital of Larissa, Dep of Medical Oncology, Larissa
  - "Metaxa's" Anticancer Hospital of Piraias, Piraeus
  - "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology, Thessaloniki

REFERENCES:
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241